CLINICAL TRIAL: NCT00331149
Title: A Randomised, Double-Blind, Double-Dummy, Parallel Group Comparison of 24 Weeks of Treatment With Ropinirole Immediate Release Tablets (REQUIP IR) or Ropinirole Prolonged Release Tablets (SK&F-101468) in Advanced Stage Parkinson's Disease Subjects Who Are Not Adequately Controlled on L-dopa.
Brief Title: A Comparison of Ropinirole Immediate Release With Ropinirole Prolonged Release in Patients With Advanced Parkinson's
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: ROP105323
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Parkinson Disease
Keywords: safety; efficacy; L-dopa; ropinirole PR; Parkinson's disease; ropinirole IR; adjunctive therapy; superiority; REQUIP; health outcomes
MeSH Terms: conditions — Parkinson Disease | interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ropinirole prolonged release
Drug: ropinirole immediate release
  Other Names: Ropinirole prolonged release

SUMMARY:
This study was designed to compare the effectiveness and tolerability of a new prolonged release formulation of ropinirole with the currently marketed immediate release formulation which is prescribed in many countries. The new prolonged release formulation allows the drug to be taken once a day rather than three times a day. This study will also evaluate the side effects of the new prolonged release formulation of ropinirole

ELIGIBILITY:
Inclusion criteria:

* Patients with a diagnosis of advanced idiopathic Parkinson's disease (according to modified Hoehn & Yahr criteria Stages II-IV) whose symptoms are not adequately controlled with L-dopa.

Exclusion criteria:

* Patients with late stage advanced Parkinson's disease with incapacitating dyskinesias on a stable dose of L-dopa.
* Current, or history of, (within the previous 3 months), significant and/or uncontrolled psychiatric, haematological, renal, hepatic, endocrinological, neurological, or cardiovascular disease or active malignancy.
* Recent history of severe dizziness or fainting on standing.
* Dementia, neurotic behaviour, crippling degenerative arthritis or limb amputations, or prior or current major psychosis.
* Recent history or current evidence of drug abuse or alcoholism.
* Use of a dopamine agonist within 4 weeks of starting the study.
* Personal or family history of an allergic reaction to ropinirole.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2006-06-20 (Actual); Primary Completion 2007-08-29 (Actual); Study Completion 2007-08-29 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with at least a 20% maintained reduction in Baseline time spent "off" at Week 24 last observation carried forward (LOCF) | Baseline (Week 0) and Week 24
  Diary cards completed by the participants was used to assess the duration of "off" and "on" periods. During the treatment period 2, 24 hour diary cards were completed by the participants (except for the Baseline period when four diary cards were completed). The participants completed diary cards on the same 2 days of each relevant week. Each 30 minute period was marked as either "off", "on" or asleep. Troublesome dyskinesias were involuntary twisting, turning movements which caused discomfort were also recorded. The general definition of "off" included a lack of mobility with or without additional features such as tremor or rigidity. The total number of hours spent both "off" and "on" or asleep were summed for the two (four for the Baseline Period) 24 hour diary cards and the amount of awake time spent "off" per 24 hour period was determined. Percentage of participants with at least a 20% maintained reduction in baseline time spent "off" at Week 24 were presented.

SECONDARY OUTCOMES:
Mean change from Baseline in percentage awake time spent "off" at Week 24 LOCF | Baseline (Week 0) and Week 24
  Diary cards completed by the Participants was used to assess the duration of "off" and "on" periods. During the Treatment Period 2 24 hour diary cards were completed by the Participants (except for the Baseline Period when four diary cards were completed). The Participants completed diary cards on the same 2 days of each relevant week. Each 30 minute period was marked as either "off", "on" or asleep. Troublesome dyskinesias were involuntary twisting, turning movements which caused discomfort were also recorded. The general definition of "off" included a lack of mobility with or without additional features such as tremor or rigidity. The total number of hours spent both "off" and "on" or asleep were summed for the two (four for the Baseline Period) 24 hour diary cards and the amount of awake time spent "off" per 24 hour period was determined. Week 0 was the baseline and change from Baseline was calculated by subtracting the baseline values from the on-treatment values.
Number of participants with a score of 'much improved' or 'very much improved' on the clinical global impression-global improvement (CGI-I) scale at Week 24 LOCF | Week 24
  The CGI-I global improvement scale allows the investigator to rate the participant's total improvement from beginning the treatment (baseline). The scale was rated as 1-7, from 1: very much improved, 2: much improved, 3: minimally improved, 4: no change, 5: minimally worse, 6: much worse and 7: very much worse. CGI global improvement scale was assessed at Week 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24 (and at early withdrawal, if applicable. Higher score indicates worsening and lower score indicates very much improvement. A participant was considered as a CGI-I responder when he/she had a score of (1) Very Much Improved or (2) Much Improved.
Mean change from baseline in the total motor score (part III) of the Unified Parkinson's Disease Rating Scale (UPDRS), with participants in an "on" state at Week 24 LOCF | Baseline (Week 0) and Week 24
  The UPDRS Part III assessed motor examination on 18-31 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms and lower score indicates less severe PD symptoms. "On" state was where PD symptoms were well controlled by the drug. Week 0 was the Baseline and change from Baseline for an individual participant was calculated by subtracting the Baseline values from the on-treatment values. Mean change from Baseline in the total motor score with participants in an "on" state was reported.
Mean change from baseline in the total motor score (part III) of the UPDRS, with participants in an "off" state at Week 24 LOCF | Baseline (Week 0) and Week 24
  The UPDRS Part III assessed motor examination on 18-31 items. Participants receive a score of 0-4 points per item. The maximum total score is 108 points. A higher score indicates more severe PD symptoms and lower score indicates less severe PD symptoms. Week 0 was the baseline and change from Baseline for an individual participant was calculated by subtracting the baseline values from the on-treatment values. Mean change from baseline in the total motor score with participants in an "off" state was reported.
Mean change from baseline in the total Activities of daily living (ADL) score (part II) of the UPDRS, with participants in an "on" state at Week 24 LOCF | Baseline (Week 0) and Week 24
  This component included items 5-17 of the UPDRS was evaluated by calculating the total score for the 13 items. Participants receive a score of 0-4 points per item and had a value ranging from 0 to 52. The maximum total score was 52. The total ADL Score of the UPDRS ranged from 0 to 52, where 0=normal/no symptoms and 52=worst possible case. Participants recorded responses in both "on" and "off" states at each visit due to the nature of questionnaire which generated ADL score at each visit. A higher score indicates more severe PD symptoms. "On" state was where PD symptoms were well controlled by the drug. Week 0 was the Baseline and change from Baseline for an individual participant was calculated by subtracting the baseline values from the on-treatment values for each state separately.
Mean change from baseline in the total ADL score (part II) of the UPDRS, with participants in an "off" state at Week 24 LOCF | Baseline (Week 0) and Week 24
  This component included items 5-17 of the UPDRS was evaluated by calculating the total score for the 13 items. Participants receive a score of 0-4 points per item and had a value ranging from 0 to 52. The maximum total score was 52. The total ADL Score of the UPDRS ranged from 0 to 52, where 0=normal/no symptoms and 52=worst possible case. Participants recorded responses in both "on" and "off" states at each visit due to the nature of questionnaire which generated ADL score at each visit. A higher score indicates more severe PD symptoms. "Off" state was where PD symptoms were not adequately controlled by the drug. Week 0 was the baseline and change from Baseline for an individual participant was calculated by subtracting the baseline values from the on-treatment values for each state separately.
Mean change from baseline in the total score (parts I-III) of the UPDRS, with participants in an "on" state at Week 24 LOCF | Baseline (Week 0) and Week 24
  The total UPDRS score was calculated by the sum of the values for each component (Part I + Part II + Part III) as determined by the physician. The UPDRS Part I scored mentation, behavior and mood and scores ranged from 0-16. The UPDRS Part II was the ADL and score ranged from 0-52. The UPDRS Part III was the Motor Examination (Total Motor Score )and scores ranged from 0-108. The total UPDRS (Part I + II + III) score ranged from 0-176 with the higher score indicating the worse condition. Tests were performed when the participant was in the "on" state of Parkinson's. Baseline was defined as Week 0 assesment. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Mean change from baseline in the total score (parts I-III) of the UPDRS, with participants in an "off" state at Week 24 LOCF | Baseline (Week 0) and Week 24
  The total UPDRS score was calculated by the sum of the values for each component (Part I + Part II + Part III) as determined by the physician. The UPDRS Part I scored mentation, behavior and mood and scores ranged from 0-16. The UPDRS Part II was the ADL and score ranged from 0-52. The UPDRS Part III was the Motor Examination (Total Motor Score)and scores ranged from 0-108. The total UPDRS (Part I + II + III) score ranged from 0-176 with the higher score indicating the worse condition. Tests were performed when the participant was in the "off" state of Parkinson's. Baseline was defined as Week 0 assessment. The change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Mean change from baseline to Week 24 LOCF in the thermometer score of the Euro-Qol 5D (EQ-5D) | Baseline (Week 0) and Week 24
  The EQ-5D was a standardized, participant-administered instrument which produced a simple descriptive profile (thermometer) and a single index value (utility) of a participant's current health status. Thermometer was a 20-cm Visual Analogue Scale (VAS) anchored at 0: worse imaginable health state and 100: best imaginable health state. Participants were required to indicate how good or bad was their health by marking a line on the scale. The point at which the line crossed the thermometer was taken as the score. Week 0 was the baseline and change from Baseline was calculated by subtracting the baseline values from the on-treatment values.
Mean change from baseline to Week 24 LOCF in the utility score of the EQ-5D | Baseline (Week 0) and Week 24
  The EQ-5D was a standardized, participant-administered instrument which produced a simple descriptive profile (thermometer) and a single index value (utility) of a participant's current health status. Utility score was computed from 5 dimensions of health: (mobility, self-care, usual activities, pain/discomfort, anxiety /depression). Each dimension comprised 3 levels (some, moderate, extreme problems), and generated a total of 243 theoretically possible health states. The Utility score was combined scores from 5 dimensions, which valued between -0.594 (representing the worse possible health) and 1 (representing the perfect health). Week 0 was the baseline and change from Baseline was calculated by subtracting the baseline values from the on-treatment values.
Mean change from Baseline in the total score of the Parkinson's Disease Sleep Scale (PDSS) at Week 24 LOCF | Baseline (Week 0) and Week 24
  The PDSS comprised of a series of 15 VAS addressing commonly reported symptoms associated with sleep disturbance in PD. The participant or caregiver completed the scale based on their experiences in the past week. Scores for each item ranged from 0 (representing the most severe) to 10 (the least severe). The maximum score for the PDSS was 150 (participant was free of all symptoms). Week 0 was the baseline and change from Baseline was calculated by subtracting the baseline values from the on-treatment values.
Mean change from Baseline in the total movement severity score of the abnormal involuntary movement scale (AIMS), with participants in an "on" state at Week 24 LOCF | Baseline (Week 0) and Week 24
  The AIMS was a 12 item, investigator performed assessment of facial and oral movements, extremity movements, trunk movements, global judgments and dental status according to predefined criteria. Items 1-10 were rated on a 5 point severity scale with 0: none to 4: severe. Items 11 and 12 were yes or no items. The AIMS total movement severity score was obtained by summing together the responses to the first seven items and ranged from 0 to 28, with higher scores representing more severe involuntary movement. The AIMS was assessed at Week 0, 12, 24. Week 0 was the baseline and change from Baseline was calculated by subtracting the baseline values from the on-treatment values.
Percentage of participants requiring re-instatement of L-dopa | Week 24
  Participants were defined as having a re-instatement of L-dopa, if at any point during the on-treatment phase (excluding down-titration), their dose of L-dopa was increased, up to, or above their baseline level. Percentage of participants requiring reinstatement of L-dopa was reported at Week 24.
Mean change from baseline in the dose of L-dopa at Week 24 LOCF | Baseline (Week 0) and Week 24
  The start and stop dates of L-Dopa medication were used to determine the dose being taken on a specific date or at an assessment. The dose recorded on the actual date of assessment was used when reporting the corresponding dose. The total daily dose of L-dopa (mg) was calculated as Unit dose per tablet (mg) * Daily Frequency * No of Tablets per administration. Mean change from baseline in the dose of L-dopa at Week 24 was reported. Week 0 was the baseline and change from Baseline was calculated by subtracting the baseline values from the on-treatment values.
Incidence of all adverse events (AE) and serious adverse events (SAE) | Up to Week 27
  Data for number of participants who presented one or more adverse events (serious or non serious) was reported. An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Number of participants who were unable to titrate weekly during the 4 week forced up titration due to poor tolerability | Up to Week 24
  There was no specific question in the CRF to capture the reason why participants were unable to titrate weekly during this period, the data on the reason for withdrawal in the CRF was thus evaluated in those participants who withdrew during the forced titration period. Data for the number of participants withdrawn (Yes/No) is presented.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (66):
- Bulgaria (2):
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (5):
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Windsor, Ontario
  - GSK Investigational Site, Québec
- Czechia (4):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Ostrava - Poruba
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
- France (6):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
- Germany (10):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Hildesheim, Lower Saxony
  - GSK Investigational Site, Westerstede, Lower Saxony
  - GSK Investigational Site, Bielefeld, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Gera, Thuringia
  - GSK Investigational Site, Berlin
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Szeged
- Italy (8):
  - GSK Investigational Site, Chieti Scalo, Abruzzo
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Grosseto, Tuscany
  - GSK Investigational Site, Lido Di Camaiore (Lucca), Tuscany
  - GSK Investigational Site, Arcugnano (VI), Veneto
- Poland (6):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Warsaw
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- South Africa (4):
  - GSK Investigational Site, Pretoria, Gauteng
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Sunninghill
- Spain (6):
  - GSK Investigational Site, Alcorcon (Madrid)
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Donostia / San Sebastian
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Sant Cugat Del Valles (Barcelona)
  - GSK Investigational Site, Seville
- Ukraine (3):
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Vinnitsa
- United Kingdom (5):
  - GSK Investigational Site, Bristol, Gloucestershire
  - GSK Investigational Site, Stoke-on-Trent, Staffordshire
  - GSK Investigational Site, Chertsey
  - GSK Investigational Site, Leigh
  - GSK Investigational Site, Oxford